CLINICAL TRIAL: NCT05954988
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation, Safety, Tolerability and Pharmacodynamic Biomarker Study of Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03) in Recently Diagnosed, Treatment Naïve Subjects With IPF
Brief Title: A Study to Evaluate LTI-03 in Newly Diagnosed Idiopathic Pulmonary Fibrosis (IPF) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rein Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: LTI-03-1002
Record Dates: First submitted 2022-05-20; First posted 2023-07-20 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sponsor, Investigator, and study personnel working on behalf of the Investigator and Sponsor will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 2.5 mg LTI-03 BID (Experimental): 2.5 mg LTI-03 BID x 14 days
  Interventions: Drug: LTI-03
- 5 mg LTI-03 BID (Experimental): 5 mg LTI-03 BID x 14 days
  Interventions: Drug: LTI-03
- Placebo (Placebo Comparator): Matching placebo BID x 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LTI-03 — Caveolin-1-Scaffolding-Protein-Derived Peptide
  Other Names: Micronized dry powder in hard 2 piece hypromellose capsules
  Arms: 2.5 mg LTI-03 BID; 5 mg LTI-03 BID
Drug: Placebo — Matching placebo
  Other Names: Micronized lactose powder in capsule
  Arms: Placebo

SUMMARY:
This study will assess the safety and tolerability of inhaled LTI-03 in treatment naïve participants with newly diagnosed IPF.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, multi-center, dose escalation, safety and tolerability study of LTI-03 or placebo administered by inhalation in participants recently diagnosed with idiopathic pulmonary fibrosis that have not received prior treatment with anti-fibrotic agents.

The study will contain 2 dose cohorts which will run sequentially.

Eligible participants will be randomized in a 3:1 ratio to either LTI-03 or placebo. Safety data will be reviewed on an ongoing basis. Enrollment in the second cohort will not begin until the Cohort 1 safety data has been reviewed.

The Treatment Period will be 14 days, with subjects self-administering study drug using a provided commercially available dry-powder inhaler.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject of age 40 years or older.
2. Willing and able to provide written informed consent.
3. Diagnosis of IPF within 3 years of Screening as confirmed by HRCT of chest or lung biopsy as defined by ATS/ERS/JRS/ALAT guideline.
4. Forced vital capacity (FVC) percent predicted ≥ 40%.
5. Diffusion capacity of the lungs for carbon monoxide (DLCO) percent predicted ≥ 30 and ≤ 80.
6. Forced expiratory volume 1 (FEV1)/FVC ≥ 0.7.

Exclusion Criteria:

1. Interstitial lung disease other than IPF.
2. Evidence of significant obstructive lung disease.
3. Current diagnosis of asthma.
4. Treatment with an approved or investigational antifibrotic therapy for IPF within 2 months of the Baseline bronchoscopy.
5. Use of N-acetyl cysteine or other supplements within 7 days prior to dosing and throughout the Treatment Period.
6. Inability to use study inhaler device appropriately.
7. Pulmonary exacerbation within 6 months prior to Screening.
8. Febrile illness within 7 days prior to dosing.
9. Participation in a clinical study or treatment with an investigational drug or device within 30 days of the Screening Visit (or 5 half-lives of the investigational agent, whichever is longer).
10. History or evidence at screening of significant renal impairment with eGFR < 30 mL/min (region specific).
11. History or evidence at screening of significant hepatic impairment with bilirubin > 3 mg/dL (> 51.3 µmol/L) and albumin < 2.8 g/dL (<28 g/L) and PT prolongation > 6 sec or INR > 2.3 (region specific).
12. Serious or active medical or psychiatric condition which, in the opinion of the Investigator, may interfere with treatment, assessment, or compliance with the protocol.
13. Vaccination within 2 weeks of start of dosing (Day 1) and throughout the Treatment Period.
14. Subject has severe progressive or uncontrolled, clinically significant disease that in the judgment of the investigator or designee renders the subject unsuitable for the study.
15. Positive urine pregnancy test in female subjects of childbearing potential as defined below.
16. Female subjects who are lactating.
17. Females of childbearing potential (FOCBP) and men with partners of childbearing potential who do not agree to use an acceptable form of contraception for the duration of study treatment and for at least 90 days after the last dose of study drug. Male subjects who do not agree to refrain from donating sperm during this same period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Shoemkaer, MD, Study Director — Lung Therapeutics
Locations (7):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
- Agaplesion Evangelisches Krankenhaus Mittelhessen, Giessen, Germany
- United Kingdom (3):
  - University of Edinburgh, Edinburgh
  - Royal Brompton Hospital, London
  - Royal Victoria Infirmary, Newcastle

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2.5 mg LTI-03 BID | 5 mg LTI-03 BID | Placebo
Started | 9 | 9 | 6
Completed | 9 | 9 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 mg LTI-03 BID | 5 mg LTI-03 BID | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 1 | 8
  >=65 years | 5 | 6 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (9.76) | 68.4 (10.79) | 71.7 (6.15) | 69.0 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 7 | 7 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 9 | 6 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 0 | 3
  United Kingdom | 3 | 2 | 3 | 8
  Germany | 3 | 4 | 2 | 10
  Australia | 1 | 2 | 1 | 3
Height [Mean (Standard Deviation); unit: cm] | 170.93 (9.270) | 169.56 (9.530) | 177.17 (7.111) | 171.98 (9.067)
Weight [Mean (Standard Deviation); unit: kg] | 84.49 (11.709) | 85.36 (25.108) | 91.45 (11.529) | 86.55 (17.446)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.869 (2.7335) | 29.364 (6.6335) | 29.330 (4.9868) | 29.170 (4.8340)
Number of Participants with Past and/or current tobacco use [Count of Participants; unit: Participants]
  Yes | 8 | 7 | 4 | 19
  No | 1 | 2 | 2 | 5
Cigarette smoking [Mean (Standard Deviation); unit: pack-years] | 18.25 (10.327) | 35.99 (22.861) | 26.88 (26.772) | 27.06 (20.331)
Diffusion capacity of the lungs for carbon monoxide (DLCO) [Mean (Standard Deviation); unit: mmol/min/kPa] | 5.123 (0.7913) | 5.020 (1.5804) | 5.354 (0.6776) | 5.143 (1.1092)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: L] | 3.214 (0.7744) | 3.318 (0.6421) | 3.085 (0.2733) | 3.221 (0.6138)
FVC percent predicted [Mean (Standard Deviation); unit: percent] | 84.789 (10.2189) | 92.111 (18.6644) | 75.617 (8.9410) | 85.242 (14.7507)
Leicester Cough Questionnaire (LCQ) Total Score [Mean (Standard Deviation); unit: units on a scale] — Range of possible total scores is 3 to 21 with higher scores indicating better quality of life related to cough. Total is sum of the mean scores for 3 domains (physical, psychological, and social). 19 questions separated into the 3 domains are answered using a 7-point Likert scale where 1 represents "all of the time" and 7 represents "none of the time".
  units on a scale | 18.19 (3.264) | 16.59 (3.236) | 16.12 (3.373) | 17.07 (3.262)
Cough Visual Analogue Scale (VAS) Score [Mean (Standard Deviation); unit: units on a scale] — Range of possible scores 0 to 100. An analogue scale with 0 = no cough and 100 = worst possible cough
  units on a scale | 29.6 (30.65) | 38.1 (21.51) | 35.3 (27.20) | 34.2 (25.75)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: Incidence of TEAEs by dose
Time Frame: 21 days (dosing x 14 days; follow up x 7 days)
Measure: Number; unit: percentage of participants
Arm/Group | 2.5 mg LTI-03 BID | 5 mg LTI-03 BID | Placebo
Number analyzed (Participants) | 9 | 9 | 6
percentage of participants
  Any TEAE | 66.7 | 77.8 | 50.0
  Any TEAE with CTCAE severity Grade 3 or higher | 0 | 0 | 0
  Any study drug-related TEAE | 22.2 | 55.6 | 16.7
  Any TEAE leading to treatment discontinuation | 0 | 0 | 0
  Any serious TEAE | 0 | 11.1 | 0
  Any TEAE leading to death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From ICF (if serious or related to protocol assessment) or Dosing Day 1 through End of Study Day 21
Arm/Group | 2.5 mg LTI-03 BID | 5 mg LTI-03 BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/9 | 0/6
Other Adverse Events (participants affected / at risk) | 6/9 | 7/9 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg LTI-03 BID (N=9) | 5 mg LTI-03 BID (N=9) | Placebo (N=6)
Post-procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg LTI-03 BID (N=9) | 5 mg LTI-03 BID (N=9) | Placebo (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 2 (2)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT05954988/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT05954988/SAP_001.pdf